CLINICAL TRIAL: NCT07247591
Title: Determination of Adductor Canal Location by USG Measurements and Cadaver Correlation
Brief Title: Adductor Canal Localization in Living and Cadaver
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yasin Usta, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2025-0249
Record Dates: First submitted 2025-09-20; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anatomy; Adductor Canal Block
Keywords: ASIS; ADDUCTOR CANAL; BLOCK

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ULTRASONOGRAPHIC PARTICIPANT GROUP: Participants will have ultrasound imaging of the adductor canal anatomy.
- Cadaver Group: Anatomical measurements and adjacencies of the adductor canal will be examined on cadavers.

SUMMARY:
The aim of this study is to define the starting and ending points of the adductor canal in adductor canal block (ACB) applications through distance measurements relative to the anterior superior iliac spine (ASIS) and the adductor tubercle. These measurements are performed using ultrasound (USG) and correlated with cadaveric data.

Key research questions addressed include:

* Can the start and end points of the adductor canal be formulated along a line drawn between the ASIS and the adductor tubercle?
* Is there a definable relationship between the block application site and anatomical landmarks such as the vastoadductor membrane (VAM), the apex of the femoral triangle, and other adjacent structures that facilitates localization?

By validating ultrasound measurements with cadaveric findings, the study aims to provide researchers with a more predictable and reliable method for determining the optimal site for adductor canal block administration.

DETAILED DESCRIPTION:
The aim of this study is to define the starting and ending points of the adductor canal (AC) in the context of adductor canal block (ACB) applications, through distance measurements related to the anterior superior iliac spine (ASIS) and adductor tubercle. These measurements are performed in two different planes: the first plane is along an imaginary line drawn between the ASIS and the femoral adductor tubercle, while the second plane is formed by the line between the ASIS and the base of the patella.

In these planes, distances were measured between the following points:

The distance between the adductor tubercle and ASIS,

The distance between ASIS and the base of the patella,

The distance between ASIS and the apex of the patella,

The distance between the midpoint of the inguinal fold and the base of the patella.

In patients, ultrasound was used to identify and mark the following anatomical points:

The apex of the iliopectineal fossa,

The first visible point of the vastoadductor membrane (VAM),

The point where the sartorius muscle ends with the intersection of the adductor longus and begins its contact with the edge of the adductor magnus point

The point where the adductor hiatus is located.

Additionally, in patients where visible, the descending genicular artery was also marked.

The position of the femoral artery in relation to the VAM (medial, middle, or lateral) was noted, as well as the location where the femoral artery intersects the adductor magnus and sartorius, and the depth from the skin to the adductor hiatus. Circumferential measurements of the thigh were also taken at these points.

Some of the data obtained was compared with anatomical measurements obtained through cadaveric dissection.

Key Research Questions

Where are the starting and ending points of the adductor canal?

Can the adductor canal be defined along a line drawn between the ASIS and the adductor tubercle?

Is there a definable relationship between the block application site and anatomical landmarks such as the vastoadductor membrane (VAM), the apex of the femoral triangle, and other adjacent structures that facilitate localization?

By validating ultrasound measurements with cadaveric findings, the study aims to provide researchers with a more predictable and reliable method for determining the optimal site for adductor canal block applications

ELIGIBILITY:
Inclusion Criteria:

ASA 1-2-3 patients

BMI <35

Ages 18-65

Those willing to participate in the study

Exclusion Criteria:

Those unwilling to participate in the study

Pregnant women

BMI >35

ASA 4-5-6 patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: He study at Etlik City Hospital will include patients who meet the following criteria: ASA classification of 1, 2, or 3, indicating individuals who are healthy or have mild to moderate systemic disease without major functional limitation; a BMI below 35 to exclude participants with obesity-related comorbidities; and an age range of 18 to 65 to ensure a broad yet controlled sample while avoiding age-related confounding factors. All participants must also provide informed consent, confirming their understanding of the study's purpose, procedures, and potential risks.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
location of the adductor canal | Perioperative/Periprocedural
  Determine the location of the adductor canal on an imaginary line drawn between the anterior superior iliac spine and the adductor tubercle..

SECONDARY OUTCOMES:
Determining the entry point for adductor canal block | Perioperative/Periprocedural
  Standardization of the entry point for adductor canal block by defining the relationship of the canal to other structures
Adductor Canal neighborhoods | Perioperative/Periprocedural
  Detection of the canal by imaging the Vasto adductor membrane
cadaver dissection | Perioperative/Periprocedural
  Determining the compatibility of the data obtained in ultrasonographic imaging with the real anatomical structures after cadaver dissection
adductor canal | Perioperative/Periprocedural
  measuring adductor canal length

CONTACTS AND LOCATIONS:
Overall Officials: Müge Çakırca, Associate Professor, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No